CLINICAL TRIAL: NCT05519280
Title: Effects of a Biopsychosocial-Spiritual Group Intervention on Quality of Life of Institutionalized Seniors With Disabilities: A Randomized Controlled Trial
Brief Title: Effects of a Biopsychosocial-Spiritual Group Intervention on Quality of Life of Institutionalized Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, The Office of Research and Development, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MOST-105-2314-B-715-002-MY3
Record Dates: First submitted 2022-08-18; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Quality of Life
Keywords: Quality of Life; Institutionalized seniors; Disabilities; Meaning in life; Biopsychosocial-Spiritual group intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the Biopsychosocial-Spiritual Group Intervention (Experimental): The experimental group received 8 sessions of weekly BPS-S group therapy for 80 minutes each.
  Interventions: Behavioral: the Biopsychosocial-Spiritual Group Intervention
- weekly general chatting activities (No Intervention): The Control group received weekly general chatting activities for 30 minutes.

INTERVENTIONS:
Behavioral: the Biopsychosocial-Spiritual Group Intervention — The Experimental group received 8 sessions of weekly BPS-S group therapy for 80 minutes each.
  Arms: the Biopsychosocial-Spiritual Group Intervention

SUMMARY:
This study aimed to evaluate the effects of a biopsychosocial-spiritual (BPS-S) Group intervention on quality of life among seniors with disabilities in long-term care residential settings.

DETAILED DESCRIPTION:
Background: Traditionally, biomedical care approach has been insufficient to meet the complex needs of older people living with multi-morbidity. Promoting whole-person wellness and better quality of life becomes a key goal of care in residential long-term care facilities. The integrative approaches composed of physio-psycho-social and spiritual components might be a viable strategy to assist older adults accept uncontrollable life changes and enhance holistic wellness.

Purpose: The study purpose was to develop and evaluate the effects of 8-week biopsychosocial-spiritual (BPS-S) group intervention versus usual care on self-perception of quality of life (QoL) and meaning in life among seniors with disability in residential care home at mid- and post-intervention, and at a 1-month follow up.

Methods: This single-blind randomized controlled trail with repeated measures design was conducted in residential long-term care facilities. Both the experimental groups (EG) and the control group (CG) received routing group activities based on their institution's schedule. Additionally, the EG received 8 sessions of weekly BPS-S group therapy for 80 minutes each. The baseline characteristics of residents with disabilities (including demographic information, length of stay in the institution and medical conditions) were collected using a data sheet, and activities of daily living of these residents were measured using the Barthel Index. To evaluate the effectiveness of the BPS-S group therapy, the primary outcomes including "participants' overall QOL" and the secondary outcome "meaning in life" were assessed at four time points: before, mid- and post- intervention and at a 1-month follow up. Quality of Life Index (QLI)-Part I and Purpose in Life (PIL) test were used to measure these outcome variables, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. being 65 years of age or older;
2. living in the institution for at least 1 month;
3. Barthel Index scores under 90;
4. no hearing, visual impairment and infectious diseases;
5. being able to follow instructions and participate in group activities.

Exclusion Criteria:

have the diagnosis of major depression.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in quality of life summary scores before intervention to 4-week post intervention. | The data were collected before the intervention to week 12: baseline, in the middle of the intervention (the fourth week), at the end of the intervention (the eighth week), and the follow-up four weeks after the intervention (the twelfth week).
  Quality of life was measured using the Chinese version of the Quality of Life Index (QLI)-Part I. It contains 33 items measuring satisfaction regarding the four domains (health and functioning, social and economic domain, psychological/spiritual wellness, and family). The QLI-Part I is a six-point satisfaction rating scale from very unsatisfied (1) to very satisfied (6). To determine the scores, each satisfaction item is recoded from -0.25 to 0.25, and both the overall and subscale scores of the QLI-Part I calculated by following step by step scoring instructions ranges from 0 to 30; highest values represent better quality of life

SECONDARY OUTCOMES:
Change in Meaning in life summary scores before intervention to 4-week post intervention. | The data were collected before the intervention to week 12: baseline, in the middle of the intervention (the fourth week), at the end of the intervention (the eighth week), and the follow-up four weeks after the intervention (the twelfth week).
  Meaning in life was measured using the Purpose in Life Test (PIL). It is a 20-item scale designed to measure the degree of perceived meaning and purpose in individual life. Each item of the original scale is rated on a seven-point scale along a continuum from one extreme feeling (0) to the opposite feeling (7). However, too many options may be difficult for older adults to make ratings, so the original seven-point scale was modified to a five-point scale in this study, with 3 representing a neutral response. Possible scores range from 20 to 100, where higher scores indicate stronger sense of meaning in life.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Heng Chen, Principal Investigator — Department of Nursing
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No